CLINICAL TRIAL: NCT06250439
Title: Effect of Peripheral VA-ECMO Flow Variations on the Pulmonary Arterial Occlusion Pressure (PAPO) in Patients With Refractory Cardiogenic Shock: the PAPO-Flow Study
Brief Title: Effect of Peripheral VA-ECMO Flow Variations on the Pulmonary Arterial Occlusion Pressure (PAPO) in Patients With Refractory Cardiogenic Shock.
Acronym: PAPO-Flow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: APHP231770
Record Dates: First submitted 2024-01-15; First posted 2024-02-09 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Cardiogenic Shock
Keywords: Cardiogenic shock; Pulmonary arterial occlusion pressure; PAOP; VA ECMO; Left ventricle unloading
MeSH Terms: conditions — Shock, Cardiogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adult patients with peripheral VA-ECMO for refractory cardiogenic shock (Experimental): Adult patients with peripheral VA-ECMO for refractory cardiogenic shock, hospitalized in medical ICU of Pitié Salpêtrière Hospital, AP-HP Paris
  Interventions: Other: ECMO-Flow variations

INTERVENTIONS:
Other: ECMO-Flow variations — The protocol unfolds in 5 steps as follows, each step lasting between 10 and 15 minutes to allow for the patient's hemodynamic adaptation. At each step, invasive and non-invasive hemodynamic evaluation is performed.
  1. The 1st step is called "100% flow": it involves recording the patient's hemodynamic measurements at the baseline, i.e., at 100% of their ECMO-VA flow, previously set by the clinician entirely independently of the study.
  2. The 2nd step is called "125% flow": the patient's ECMO-VA flow is increased to 125% of the initial flow.
  3. The 3rd step is called "150% flow": the patient's ECMO-VA flow is increased to 150% of the initial flow.
  4. The 4th step is called "175% flow": the patient's ECMO-VA flow is increased to 175% of the initial flow.
  5. The 5th and final step is called "200% flow": the patient's ECMO-VA flow is increased to 200% of the initial flow.

SUMMARY:
This study focuses on a population of adult patients placed under peripheral Veno-Arterial Extracorporeal Membrane Oxygenation (VA-ECMO) for refractory cardiogenic shock. Cardiogenic shock, primarily caused by myocardial infarction, is associated with a high mortality rate that remains around 50%, despite advancements in the field of coronary reperfusion. VA-ECMO is a rapidly growing cardiac support technique worldwide. Its goal is to improve peripheral organ perfusion even as myocardial damage continues, thereby enhancing the prognosis of patients with severe multiorgan failure. VA-ECMO is a temporary cardio-respiratory support technique based on the principle of extracorporeal circulation. However, patients under VA-ECMO are at risk of experiencing various complications, including infectious, thromboembolic, hemorrhagic complications, or malfunctions of the ECMO machine itself, with the incidence increasing with the duration of assistance.

Numerous authors and scientific reviews highlight the increased risk of Acute Pulmonary Edema (APE) in patients under peripheral VA-ECMO, attributing it to the elevation of afterload induced by retrograde arterial reinfusion against the residual native blood flow, hypothetically leading to an increase in Pulmonary Artery Occlusion Pressure (PAOP). This phenomenon is presumed to intensify as the VA-ECMO reinfusion rate increases. Furthermore, APE under ECMO-VA represents a turning point in the patient's course. Brechot et al. demonstrated that patients who developed APE under VA-ECMO had a prolonged ECMO duration, a higher reliance on mechanical ventilation, an extended stay in critical care, and a higher mortality rate compared to patients who had previously undergone a left ventricular unloading technique (aimed at reducing PAOP and the risk of APE).

However, until now, no physiological study has assessed the specific effect of the variation in peripheral VA-ECMO flow on the change in PAOP during a dedicated protocol. It is with the aim of addressing this question that the investigators are considering the PAPO-Flow study.

DETAILED DESCRIPTION:
Cardiogenic shock is the most severe form of heart failure. It is characterized by acute and profound myocardial contractile dysfunction, leading to a severe decrease in cardiac index (<2.2 L/min) associated with signs of peripheral hypoperfusion. In its most severe forms, the impairment of cardiac contractile function is associated with an intense systemic inflammatory response syndrome (SIRS), leading to multiorgan failure and patient death. The mortality rate for patients in this situation is very high, approaching 50%.

Over the last decades, mechanical circulatory support techniques have gained interest, and their use in patients with cardiogenic shock refractory to medical treatments has significantly increased worldwide. Peripheral Veno-Arterial Extracorporeal Membrane Oxygenation (VA-ECMO) is the main temporary cardiac support technique used to maintain sufficient blood perfusion to the organs while awaiting myocardial recovery or heart transplantation. Its principle involves draining venous blood near the right atrium through a cannula inserted percutaneously or surgically into the patient's femoral vein. The venous blood is then reinfused after extracorporeal oxygenation into the descending aorta, countering the natural blood flow, via another cannula inserted into the femoral artery.

It has been postulated that the retrograde blood reinfusion by ECMO could increase cardiac afterload, enhance cardiac workload, and consequently reduce its own perfusion and recovery capabilities. Additionally, it has been suggested that, through this same effect, Pulmonary Artery Occlusion Pressure (PAOP) could rise, leading to acute pulmonary edema (APE), found in 30% of patients under peripheral ECMO. This, in turn, worsens the patient's tissue oxygenation and, ultimately, prognosis. According to this principle, this effect would amplify as the ECMO flow, set by the clinician, increases.

Several authors have written about this phenomenon, considering these hypothetical physiological considerations. However, to date, no prospective study has confirmed that the sequential increase in ECMO flow leads to a correlated elevation in PAOP in patients placed under peripheral VA-ECMO for refractory cardiogenic shock. Moreover, several factors may oppose this principle.

Firstly, as VA-ECMO retrogradely injects blood into the aorta via the arterial route, it simultaneously unloads the right cardiac chambers by an equivalent amount (in liters/minute) and reduces cardiac preload. Consequently, the filling of the left cardiac chambers and the left ventricular end-diastolic volume, both determinants of PAOP, are diminished. Secondly, arterial reinfusion by peripheral ECMO occurs more than 30 cm from the aortic valve, and its effect on cardiac afterload may be minimal, especially in patients with residual cardiac ejection. Finally, patients in cardiogenic shock under ECMO often present severe circulatory insufficiency, leading to significant volume expansion. They may have a markedly positive sodium-water balance, which alone could explain the elevation of PAOP and the occurrence of APE independently of the ECMO effect.

Thus, to date, the investigators do not have enough scientific evidence to certify that the variation in peripheral VA-ECMO flow alone induces an increase in PAOP in patients with refractory cardiogenic shock under peripheral VA-ECMO It is with the aim of addressing this question that the investigators are considering the PAPO-Flow study.

All eligible patients from the medical intensive care unit of the Pitié-Salpêtrière Hospital Group will be included after verification of inclusion and exclusion criteria by the investigator, explanation of the study, and provision of the information sheet. After allowing the patient a necessary reflection period to make their decision, written and voluntary consent will be obtained. If the patient is not able to understand the information or express written consent at the time of inclusion, information and consent will be obtained from their relative. Emergency inclusion will be possible if the patient is unable to understand the information or express consent, and if contacting a relative is not possible at the time of patient inclusion. Patient information and consent collection to continue participation will be sought as soon as their condition allows.

Patient demographic data, clinical data including medical history, vital signs, fluid and sodium balance, and administered treatments will be collected at the time of patient inclusion.

The protocol unfolds in 5 steps as follows, each step lasting between 10 and 15 minutes to allow for the patient's hemodynamic adaptation. At each step, invasive and non-invasive hemodynamic evaluation is performed.

1. The 1st step is called "100% flow": it involves recording the patient's hemodynamic measurements at the baseline, i.e., at 100% of their ECMO-VA flow, previously set by the clinician entirely independently of the study.
2. The 2nd step is called "125% flow": the patient's ECMO-VA flow is increased to 125% of the initial flow.
3. The 3rd step is called "150% flow": the patient's ECMO-VA flow is increased to 150% of the initial flow.
4. The 4th step is called "175% flow": the patient's ECMO-VA flow is increased to 175% of the initial flow.
5. The 5th and final step is called "200% flow": the patient's ECMO-VA flow is increased to 200% of the initial flow.

At the end of the protocol, the ECMO flow is returned to its initial value (100%) without posing any risk to the patient.

At each step of the protocol, hemodynamic tolerance is assessed through continuous monitoring of vital signs on the patient's scope by the study investigators. The protocol is interrupted in case of poor patient tolerance, and the ECMO-VA flow is immediately returned to its initial value. The patient then continues their follow-up as planned.

ELIGIBILITY:
Inclusion Criteria:

Major patient hospitalized in the medical intensive care unit at Pitié-Salpêtrière Hospital, under peripheral VA-ECMO for refractory cardiogenic shock and already equipped with a previously placed pulmonary arterial catheter before the study.

The patient must be deemed "stabilized under ECMO" by one of the study investigators so that variations in VA-ECMO flow can be tolerated.

Inclusion criteria are as follows:

1. Patient aged 18 years or older.
2. Patient hospitalized in the medical intensive care unit at Pitié-Salpêtrière Hospital.
3. Patient on peripheral veno-arterial ECMO (Extracorporeal membrane oxygenation).
4. Patient already equipped with a Swan-Ganz pulmonary arterial catheter and a radial arterial catheter (right or left) installed as part of the care.
5. Patient judged stabilized under ECMO by the study investigators to tolerate variations in VA-ECMO flow (stabilization of catecholamine levels in the preceding hours, absence of severe pulmonary function impairment, no need for a transfusion of blood products within the following 2 hours).
6. Patient or patient's representative (if the patient is not able to express themselves), having received informed information about the study, and whose written and voluntary consent has been obtained. Emergency inclusion will be possible in case the patient and their representative are unable to be informed and/or provide consent for the patient's inclusion.
7. Patient affiliated with or entitled to a social security scheme (excluding State Medical Assistance)

Exclusion Criteria:

1. SAPS-II Score > 90 (Simplified Acute Physiology Score (SAPS-II)) at inclusion (calculated as part of the care).
2. Patient unable to tolerate variations in VA-ECMO flow due to ongoing major hemodynamic instability.
3. Patient under legal protection measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2025-01-13 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
PAPO variation | during 1 day after inclusion
  Measurement of the variation in occluded pulmonary arterial pressure (PAOP in mmHg) using the pulmonary arterial catheter during different stages of peripheral VA-ECMO flow variation.
  The variation in PAOP (ΔPAOP) is the calculated difference between the PAOP measured at the end of the protocol (PAOP200%) and that measured at the beginning of the protocol (PAOP100%), estimated as a percentage according to the following formula:
  ΔPAOP(%) = (PAOP200% - PAOP100%) / PAOP200% × 100 In accordance with literature, a 20% variation in PAOP between the two flow rates will be considered significant.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de réanimation médicale, Hôpital Pitié-Salpêtrière,, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.